CLINICAL TRIAL: NCT07114978
Title: Prognostic Value of the Left Ventricular Outflow Tract Velocity-time Integral in Predicting In-hospital Outcomes in Patients Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Prognostic Value of the LVOT VTI in STEMI Patients Undergoing PPCI
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Khaled Ahmed Abdel Rahman, Principal Investigator, Assiut University
Other Study IDs: LVOT VTI in STEMI
Record Dates: First submitted 2025-07-21; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: LVOT VTI; STEMI - ST Elevation Myocardial Infarction (MI); Primary Percutaneous Coronary Intervention
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: LVOT VTI < 15 cm
  Interventions: Device: Echocardiography
- Group B: LVOT VTI ≥ 15 cm
  Interventions: Device: Echocardiography

INTERVENTIONS:
Device: Echocardiography — simple, bedsided, non-invasive

SUMMARY:
* To determine whether LVOT VTI < 15 cm predicts the development of in-hospital cardiogenic shock or need for vasopressors in STEMI patients undergoing primary PCI.
* To assess association of LVOT VTI with other adverse outcomes (in-hospital death, heart failure, arrhythmias, need for mechanical ventilation, prolonged hospital stay).

DETAILED DESCRIPTION:
ST-elevation myocardial infarction (STEMI) remains a leading cause of cardiovascular mortality globally, with an estimated incidence of 50-100 cases per 100,000 person and accounting for nearly 30% of acute coronary syndrome (ACS) presentations. Despite advances in reperfusion therapy, in-hospital complications such as cardiogenic shock (CS) and acute heart failure (HF) continue to affect 5-15% of STEMI patients, with CS-associated mortality exceeding 40%.

Primary percutaneous coronary intervention (PCI) is the standard of care in STEMI patients, but also early identification of high-risk patients is crucial to improving outcomes.

Echocardiographic evaluation of left ventricular outflow tract velocity-time integral (LVOT VTI) has gained attention as a dynamic, bedside echocardiographic parameter that reflects stroke volume (SV) and cardiac output (CO). Several studies in critically ill patients and those with heart failure have shown that low LVOT VTI values (<15 cm) are associated with impaired cardiac output and adverse outcomes, including hypotension, vasopressor requirement, and increased mortality. Moreover, in cardiogenic shock, LVOT VTI has demonstrated superior prognostic accuracy compared to conventional measures such as left ventricular ejection fraction (LVEF).

Despite this growing evidence, the prognostic role of LVOT VTI in STEMI patients remains under-investigated. Since STEMI-related LV dysfunction directly impacts stroke volume, LVOT VTI may offer an early, non-invasive indicator of impending hemodynamic deterioration ـــ potentially before clinical signs become evident. Early identification of those high-risk patients mandates careful hemodynamic monitoring and rapid management of any deterioration.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years), diagnosed with acute STEMI according to current ESC guidelines(3) and undergoing primary PCI within 24 hours of symptom onset.
2. Patients undergo transthoracic echocardiography within 24 hours of admission.

Exclusion Criteria:

1. Presence of significant aortic valve disease (e.g., severe aortic stenosis or regurgitation).
2. LVOT obstruction or hypertrophic cardiomyopathy.
3. Poor echocardiographic window.
4. Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients (aged ≥18 years) diagnosed with acute ST-segment elevation myocardial infarction (STEMI) who are admitted to Assiut University Hospital - Cardiology Department and undergo primary percutaneous coronary intervention (PCI) within 24 hours of symptom onset.
  Eligible patients will receive transthoracic echocardiography (TTE) including LVOT VTI measurement within the first 24 hours of admission as part of their routine clinical evaluation.
  Patients will be prospectively enrolled and followed during hospitalization for the occurrence of adverse in-hospital events such as cardiogenic shock, heart failure, arrhythmias, mechanical ventilation, or in-hospital mortality.
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of cardiogenic shock in patients with LVOT VTI < 15 cm | Through hospital stay (up to 3 days)
  Cardiogenic shock defined per ESC 2023 criteria (SBP <90 mmHg for ≥30 minutes plus signs of hypoperfusion, or need for vasopressors/inotropic support). Assessed during hospital stay in relation to baseline LVOT VTI.
  Unit of Measure: Percentage of patients (%)

SECONDARY OUTCOMES:
Incidence of acute heart failure in patients with LVOT VTI < 15 cm | Through hospital stay (up to 3 days)
  Defined by signs/symptoms requiring intravenous diuretics or ventilatory support, assessed during hospital stay.
  Unit of Measure: Percentage of patients (%)
Incidence of ventricular arrhythmias in patients with LVOT VTI < 15 cm | Through hospital stay (up to 3 days)
  Occurrence of sustained VT or VF requiring intervention, assessed through hospital stay.
  Unit of Measure: Percentage of patients (%)
Need for mechanical ventilation in patients with LVOT VTI < 15 cm | Through hospital stay (up to 3 days)
  Use of invasive or non-invasive mechanical ventilatory support during hospital stay.
  Unit of Measure: Percentage of patients (%)
Length of hospital stay | Through study completion (an average 1 year )
  Number of days from admission to discharge. Unit of Measure: Days

CONTACTS AND LOCATIONS:
Overall Officials: Hosam Hasan Ali Mohamed, Professor, Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aboelkasem Ali Mousa M, Abdelsabour Abdallah M, Shamseddin Mohammad H, Ahmad Aly Youssef A. Early predictors of left ventricular remodeling after primary percutaneous coronary intervention. Egypt Heart J. 2018 Dec;70(4):403-407. doi: 10.1016/j.ehj.2018.05.003. Epub 2018 Aug 24. No abstract available. PMID 30591763
- [Background] Machado GP, Telo GH, de Araujo GN, da Rosa Barbato JP, Amon A, Martins A, Nassif M, Azevedo W, da Silveira AD, Scolari FL, Pagnoncelli A, Goncalves SC, Truesdell AG, Wainstein R, Wainstein M. A combination of left ventricular outflow tract velocity time integral and lung ultrasound to predict mortality in ST elevation myocardial infarction. Intern Emerg Med. 2024 Nov;19(8):2167-2176. doi: 10.1007/s11739-024-03719-z. Epub 2024 Jul 24. PMID 39044051
- [Background] Ochagavia A, Palomo-Lopez N, Fraile V, Zapata L. Hemodynamic monitoring and echocardiographic evaluation in cardiogenic shock. Med Intensiva (Engl Ed). 2024 Oct;48(10):602-613. doi: 10.1016/j.medine.2024.07.001. Epub 2024 Aug 2. PMID 39097480
- [Background] Gentile F, Buoncristiani F, Sciarrone P, Bazan L, Panichella G, Gasparini S, Chubuchny V, Taddei C, Poggianti E, Fabiani I, Petersen C, Lancellotti P, Passino C, Emdin M, Giannoni A. Left ventricular outflow tract velocity-time integral improves outcome prediction in patients with secondary mitral regurgitation. Int J Cardiol. 2023 Dec 1;392:131272. doi: 10.1016/j.ijcard.2023.131272. Epub 2023 Aug 19. PMID 37604287
- [Background] Yuriditsky E, Mitchell OJ, Sibley RA, Xia Y, Sista AK, Zhong J, Moore WH, Amoroso NE, Goldenberg RM, Smith DE, Jamin C, Brosnahan SB, Maldonado TS, Horowitz JM. Low left ventricular outflow tract velocity time integral is associated with poor outcomes in acute pulmonary embolism. Vasc Med. 2020 Apr;25(2):133-140. doi: 10.1177/1358863X19880268. Epub 2019 Nov 10. PMID 31709912
- [Background] Omote K, Nagai T, Iwano H, Tsujinaga S, Kamiya K, Aikawa T, Konishi T, Sato T, Kato Y, Komoriyama H, Kobayashi Y, Yamamoto K, Yoshikawa T, Saito Y, Anzai T. Left ventricular outflow tract velocity time integral in hospitalized heart failure with preserved ejection fraction. ESC Heart Fail. 2020 Feb;7(1):167-175. doi: 10.1002/ehf2.12541. Epub 2019 Dec 18. PMID 31851433
- [Background] Cheong I, Castro VO, Gomez RA, Merlo PM, Tamagnone FM. A modified subcostal view: a novel method for measuring the LVOT VTI. J Ultrasound. 2023 Jun;26(2):429-434. doi: 10.1007/s40477-022-00671-6. Epub 2022 Apr 21. PMID 35449385
- [Background] Byrne RA, Rossello X, Coughlan JJ, Barbato E, Berry C, Chieffo A, Claeys MJ, Dan GA, Dweck MR, Galbraith M, Gilard M, Hinterbuchner L, Jankowska EA, Juni P, Kimura T, Kunadian V, Leosdottir M, Lorusso R, Pedretti RFE, Rigopoulos AG, Rubini Gimenez M, Thiele H, Vranckx P, Wassmann S, Wenger NK, Ibanez B; ESC Scientific Document Group. 2023 ESC Guidelines for the management of acute coronary syndromes. Eur Heart J. 2023 Oct 12;44(38):3720-3826. doi: 10.1093/eurheartj/ehad191. No abstract available. PMID 37622654
- [Background] Thiele H, Ohman EM, de Waha-Thiele S, Zeymer U, Desch S. Management of cardiogenic shock complicating myocardial infarction: an update 2019. Eur Heart J. 2019 Aug 21;40(32):2671-2683. doi: 10.1093/eurheartj/ehz363. PMID 31274157
- [Background] Vogel B, Claessen BE, Arnold SV, Chan D, Cohen DJ, Giannitsis E, Gibson CM, Goto S, Katus HA, Kerneis M, Kimura T, Kunadian V, Pinto DS, Shiomi H, Spertus JA, Steg PG, Mehran R. ST-segment elevation myocardial infarction. Nat Rev Dis Primers. 2019 Jun 6;5(1):39. doi: 10.1038/s41572-019-0090-3. PMID 31171787
- See also: Lüsebrink, E., Binzenhöfer, L., Adamo, M., Lorusso, R., Mebazaa, A., Morrow, D. A., Price, S., Jentzer, J. C., Brodie, D., Combes, A., & Thiele, H. (2024). Cardiogenic shock. Lancet (London, England), 404(10466), 2006-2020. — https://pubmed.ncbi.nlm.nih.gov/39550175/